CLINICAL TRIAL: NCT04111614
Title: A PHASE 1, RANDOMIZED, OPEN LABEL, 2 PERIOD, CROSS OVER, SINGLE DOSE STUDY TO DEMONSTRATE THE AREA UNDER THE CURVE EQUIVALENCE BETWEEN TOFACITINIB ORAL SOLUTION FORMULATION AND TABLET FORMULATION UNDER FASTED CONDITION IN HEALTHY PARTICIPANTS
Brief Title: A Study to Demonstrate the Equivalence of the Tofacitinib Oral Solution to the Tablet Formulation in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A3921354
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Single dose of 5 mL tofacitinib oral solution on Day 1 of Period 1 and Singe dose of 5 mg tofacitinib tablet on Day 1 of Period 2
  Interventions: Drug: Tofacitinib tablet; Drug: Tofacitinib Oral Solution
- Arm 2 (Experimental): Single dose of 5 mg tofacitinib tablet on Day 1 of Period 1 and Singe dose of 5 mL tofacitinib oral solution on Day 1 of Period 2
  Interventions: Drug: Tofacitinib tablet; Drug: Tofacitinib Oral Solution

INTERVENTIONS:
Drug: Tofacitinib tablet — Single dose of tofacitinib 5 mg tablet
Drug: Tofacitinib Oral Solution — Single 5 mL dose of tofacitinib oral solution (1 mg/mL)

SUMMARY:
This is a Phase 1, randomized, open label, 2 period, 2 sequence, cross over, single dose study to evaluate the AUC equivalence, and safety of tofacitinib 5 mL oral solution (1 mg/mL) and 5 mg tablet in healthy participants. Participants will be randomized to 1 of the 2 treatment sequences. A total of approximately 12 healthy male and/or female (non-childbearing potential) participants will be enrolled in the study so that approximately 6 participants will be enrolled in each treatment sequence. Each treatment sequence will consist of 2 periods. In both sequences, participants will remain in the CRU for a total of 5 days and 4 nights (including Period 1 and Period 2).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of non childbearing potential must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).
* Male and female participants of non-childbearing potential who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, blood pressure (BP), pulse rate, oral temperature, and 12 lead electrocardiogram (ECG).
* Body mass index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight greater than 50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic (including alcoholic liver disease, nonalcoholic steatohepatitis (NASH), autoimmune hepatitis, and hereditary liver diseases), psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically significant infections within the past 3 months prior to the baseline visit (for example, those requiring hospitalization or parenteral antibiotics, or as judged by the investigator), evidence of any infection within the past 7 days prior to the baseline visit, history of disseminated herpes simplex infection or recurrent (>1 episode) herpes zoster or disseminated herpes zoster.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* Malignancy or a history of malignancy, with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* A positive urine drug test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
AUCinf for tofacitinib oral solution and tofacitinib tablet | 24 hrs after study drug administration in Period 1 and Period 2
  Area under the curve from time zero to extrapolated infinite time for both oral solution and tofacitinib.
AUClast for tofacitinib oral solution and tofacitinib tablet | 24 hrs after study drug administration in Period 1 and Period 2
  Area under the plasma concentration time curve from 0 to time of the last measurement of both the tofacitinib oral solution and tofacitinib tablet.

SECONDARY OUTCOMES:
Cmax for tofacitinib oral solution and tofacitinib tablet | 24 hrs after study drug administration in Period 1 and Period 2
  Maximum observed plasma concentration for tofacitinib oral solution and tofacitinib tablet
Number of subjects with adverse events (AEs). | Screening to up to 28-35 days after the last dose of study medication in Period 2.
  Number of subjects with adverse events (AEs).
Number of subjects with laboratory tests findings of potential clinical importance | Screening through Day 2 of Period 2
  Number of subjects with laboratory tests findings of potential clinical importance
Number of subjects with clinically significant abnormal vital signs | Screening through Day 2 of Period 2
  Number of subjects with clinically significant abnormal vital signs
Number of subjects with clinically significant physical examination findings | Screening to Day 2 of Period 2
  Number of subjects with clinically significant physical examination findings.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Chang C, Vong C, Wang X, Hazra A, Diehl A, Nicholas T, Mukherjee A. Tofacitinib pharmacokinetics in children and adolescents with juvenile idiopathic arthritis. CPT Pharmacometrics Syst Pharmacol. 2024 Apr;13(4):599-611. doi: 10.1002/psp4.13104. Epub 2024 Jan 31. PMID 38298058
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921354